CLINICAL TRIAL: NCT00113165
Title: A Multicenter, Double-Blind, Randomized, Parallel-group Evaluation of LAMICTAL Extended-release Adjunctive Therapy in Subjects With Partial Seizures
Brief Title: Study Evaluating LAMICTAL Extended-Release Therapy Added To Current Seizure Treatments In Patients With Partial Seizures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LAM100034
Record Dates: First submitted 2005-06-06; First posted 2005-06-07 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-12

CONDITIONS: Epilepsy; Epilepsy, Partial
Keywords: partial seizures; Epilepsy; antiepileptic drugs; anticonvulsants; LAMICTAL; seizures; lamotrigine
MeSH Terms: conditions — Epilepsy; Epilepsies, Partial; Seizures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: LAMICTAL extended-release

SUMMARY:
This study is being conducted to compare the efficacy and safety of LAMICTAL (lamotrigine) extended-release with placebo in the treatment of partial seizures. LAMICTAL extended-release is an investigational drug. Placebo tablets look like LAMICTAL extended-release tablets but do not contain active medication. In this study, LAMICTAL extended-release or placebo tablets will be added to current seizure treatments.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of epilepsy with partial seizures for more than 24 weeks.
* Must experience at least 8 partial seizures during an 8-week Baseline Phase.
* Must currently be receiving treatment with a stable regimen of one or two antiepileptic drugs for at least four weeks.
* Patient or parent/caregiver must be willing and able to maintain a written daily seizure diary.

Exclusion criteria:

* Previous treatment with lamotrigine.
* Exhibits any primary generalized seizures.
* Receiving treatment with felbamate or currently following the ketogenic diet.
* Pregnant, breastfeeding, or planning to become pregnant.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2004-10; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
The efficacy of LAMICTAL extended-release therapy will be measured by the percentage change from Baseline in partial seizure frequency during the double-blind treatment phase. | 24 Weeks

SECONDARY OUTCOMES:
Reduction in partial seizure frequency during portions of double-blind phase (=25%,=50%,=75%,100%). Time to 50% reduction in partial seizure frequency. Adverse events. Weight change. Health outcomes questionnaires. Population Pharmacokinetics | 24 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (119):
- United States (63):
  - GSK Investigational Site, Anniston, Alabama
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Northport, Alabama
  - GSK Investigational Site, Tuscaloosa, Alabama
  - GSK Investigational Site, Mesa, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Scottsdale, Arizona
  - GSK Investigational Site, Sun City, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Newport Beach, California
  - GSK Investigational Site, Santa Monica, California
  - GSK Investigational Site, Sepuldeva, California
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Hollywood, Florida
  - GSK Investigational Site, Maitland, Florida
  - GSK Investigational Site, Ocala, Florida
  - GSK Investigational Site, Tallahassee, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Augusta, Georgia
  - GSK Investigational Site, Austell, Georgia
  - GSK Investigational Site, Savannah, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Flossmoor, Illinois
  - GSK Investigational Site, Springfield, Illinois
  - GSK Investigational Site, Des Moines, Iowa
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Crestview Hills, Kentucky
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Grand Rapids, Michigan
  - GSK Investigational Site, Traverse City, Michigan
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Chesterfield, Missouri
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Edison, New Jersey
  - GSK Investigational Site, West Orange, New Jersey
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Plainview, New York
  - GSK Investigational Site, Asheville, North Carolina
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Greenville, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Cheswick, Pennsylvania
  - GSK Investigational Site, Greensburg, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Galveston, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Wichita Falls, Texas
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Seattle, Washington
  - GSK Investigational Site, Milwaukee, Wisconsin
- GSK Investigational Site, Capital Federal, Buenos Aires, Argentina
- Brazil (2):
  - GSK Investigational Site, Curitiba, Paraná
  - GSK Investigational Site, Campinas, São Paulo
- GSK Investigational Site, Santiago, Región Metro de Santiago, Chile
- Germany (40):
  - GSK Investigational Site, Singen, Baden-Wurttemberg
  - GSK Investigational Site, Ulm, Baden-Wurttemberg
  - GSK Investigational Site, Alzenau in Unterfranken, Bavaria
  - GSK Investigational Site, Bamberg, Bavaria
  - GSK Investigational Site, Fürth, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Neuötting, Bavaria
  - GSK Investigational Site, Straubing, Bavaria
  - GSK Investigational Site, Unterhaching, Bavaria
  - GSK Investigational Site, Würzburg, Bavaria
  - GSK Investigational Site, Bernau bei Berlin, Brandenburg
  - GSK Investigational Site, Ludwigsfelde, Brandenburg
  - GSK Investigational Site, Hamburg, Hamburg
  - GSK Investigational Site, Bad Homburg, Hesse
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Giessen, Hesse
  - GSK Investigational Site, Bückeburg, Lower Saxony
  - GSK Investigational Site, Göttingen, Lower Saxony
  - GSK Investigational Site, Osnabrück, Lower Saxony
  - GSK Investigational Site, Wismar, Mecklenburg-Vorpommern
  - GSK Investigational Site, Baesweiler, North Rhine-Westphalia
  - GSK Investigational Site, Bochum, North Rhine-Westphalia
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Hattingen, North Rhine-Westphalia
  - GSK Investigational Site, Mönchengladbach, North Rhine-Westphalia
  - GSK Investigational Site, Münster, North Rhine-Westphalia
  - GSK Investigational Site, Limburgerhof, Rhineland-Palatinate
  - GSK Investigational Site, Chemnitz, Saxony
  - GSK Investigational Site, Flöha, Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Radeberg, Saxony
  - GSK Investigational Site, Bernburg, Saxony-Anhalt
  - GSK Investigational Site, Halle, Saxony-Anhalt
  - GSK Investigational Site, Magdeburg, Saxony-Anhalt
  - GSK Investigational Site, Naumburg, Saxony-Anhalt
  - GSK Investigational Site, Kiel, Schleswig-Holstein
  - GSK Investigational Site, Berlin, State of Berlin
  - GSK Investigational Site, Jena, Thuringia
  - GSK Investigational Site, Jena-Lobeda, Thuringia
- India (3):
  - GSK Investigational Site, Hyderabad, Andhra Pradesh
  - GSK Investigational Site, Lucknow
  - GSK Investigational Site, New Delhi
- Puerto Rico (2):
  - GSK Investigational Site, San Germán, Puerto Rico
  - GSK Investigational Site, San Juan, Puerto Rico
- Russia (3):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Yekaterinburg
- GSK Investigational Site, Seoul, South Korea
- Ukraine (3):
  - GSK Investigational Site, Kharkiv
  - GSK Investigational Site, Kyiv
  - GSK Investigational Site, Lviv

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Naritoku DK, Warnock CR, Messenheimer JA, Borgohain R, Evers S, Guekht AB, Karlov VA, Lee BI, Pohl LR. Lamotrigine extended-release as adjunctive therapy for partial seizures. Neurology. 2007 Oct 16;69(16):1610-8. doi: 10.1212/01.wnl.0000277698.33743.8b. PMID 17938371
- [Derived] van Dijkman SC, de Jager NCB, Rauwe WM, Danhof M, Della Pasqua O. Effect of Age-Related Factors on the Pharmacokinetics of Lamotrigine and Potential Implications for Maintenance Dose Optimisation in Future Clinical Trials. Clin Pharmacokinet. 2018 Aug;57(8):1039-1053. doi: 10.1007/s40262-017-0614-5. PMID 29363050
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: LAM100034 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: LAM100034 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: LAM100034 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: LAM100034 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: LAM100034 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: LAM100034 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: LAM100034 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register